CLINICAL TRIAL: NCT00289523
Title: Biomarkers for Rapid Identification of Treatment Effectiveness in Major Depression (BRITE-MD), a Prospective, Randomized, Multi-center Study to Determine the Efficacy of Selected EEG and Genotype Biomarkers for Predicting Response to Antidepressant Therapy With Escitalopram, Bupropion XL, or a Combination Treatment Regimen.
Brief Title: EEG Biomarkers for Predicting Response to Antidepressant Therapy
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 227
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2010-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder, Depressive Disorder, Unipolar Depression, Antidepressants, Electroencephalography
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Escitalopram
- Bupropion XL
- Combination Therapy: Escitalopram and Bupropion XL

SUMMARY:
The purpose of this study is to evaluate the potential early EEG predictors of an individual's response to treatment with antidepressant medications.

Objectives:

* Prospectively confirm accuracy of current EEG biomarker algorithm
* Determine preferred clinical intervention for subjects with negative indicator
* Identify predictors of worsening suicide ideation

DETAILED DESCRIPTION:
According to recent clinical studies sponsored by the NIH, fewer than half of subjects diagnosed with a major depressive episode respond to the first trial of an antidepressant medication. While the majority of subjects eventually respond to treatment with an antidepressant, failure with the first line medication puts subjects at increased risk for never receiving adequate treatment of their depression.

Several lines of reasoning support the rationale for further investigating EEG as a means of predicting response and resistance to antidepressants. Prior studies suggest that changes in neuronal activity in the anterior cingulate and prefrontal regions are related to depression and that changes in brain response to treatment may also produce alterations that can be detected by recoding frontal EEG activity.

In this protocol, we proposed to identify possible neurophysiologic indicators of treatment outcome in depression, particularly indicators of brain response that appear early (within 7 days) during treatment with antidepressants. We will test whether quantitative EEG (QEEG) biomarkers can be reliably associated with response or non-response to treatment with antidepressant medications, using both monotherapy and combination drug treatments.

Comparison(s):

Selecting the best treatment for subjects with resistance to an initial antidepressant poses a considerable challenge for clinicians. The most widely prescribed antidepressants usually require 4-6 weeks of therapeutic dosing before a marked clinical improvement in symptoms is observed. Therefore, determining the optimal regimen can take several weeks or months for subjects who are resistant to the first line antidepressant. A tool for predicting eventual clinical response to antidepressants could help inform and accelerate the process of identifying the most efficacious treatment option for a given subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of Major Depressive Disorder

Exclusion Criteria:

* Subject is suffering from cognitive, bipolar, or psychotic disorder
* Subject has had a course of ECT within the past six months
* Subject has any known contraindication for use of any of the study drugs
* Subject has a known drug dependency or substance abuse within the past six mon ths
* Subject is currently pregnant or not using a medically acceptable means of birth control

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 375 subjects with major depressive disorder (MDD) between the ages of 18 - 75 with no other primary neuropsychiatric illnesses were recruited from the population presenting for ongoing treatment in a primary care clinic, or for depression in a psychiatric clinic at each site.
Sampling Method: Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
1. To confirm prospectively the accuracy of an EEG biomarker as a leading indicator of SSRI antidepressant treatment response; | 8 weeks
  2. To identify the optimal positive and negative indicators of response to initial treatment with an SSRI; 3. To determine the preferred clinical intervention to perform following an initial negative treatment response indicator;

SECONDARY OUTCOMES:
1. To confirm prospectively the accuracy of an EEG biomarker as a leading indicator of remission; | 8 weeks
  2. To explore the relationship between EEG and genetic biomarkers as predictors of treatment response and remission; 3. To determine if certain baseline EEG values or changes early in the course of treatment may predict the emergence of worsening suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F Leuchter, M.D., Principal Investigator — University of California, Los Angeles-Westwood
Locations (10):
- United States (10):
  - University of California, Los Angeles-Westwood, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, Los Angeles-Harbor, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas
  - Baylor University College of Medicine, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas

REFERENCES:
- [Result] Leuchter AF, Cook IA, Marangell LB, Gilmer WS, Burgoyne KS, Howland RH, Trivedi MH, Zisook S, Jain R, McCracken JT, Fava M, Iosifescu D, Greenwald S. Comparative effectiveness of biomarkers and clinical indicators for predicting outcomes of SSRI treatment in Major Depressive Disorder: results of the BRITE-MD study. Psychiatry Res. 2009 Sep 30;169(2):124-31. doi: 10.1016/j.psychres.2009.06.004. Epub 2009 Aug 27. PMID 19712979
- [Result] Leuchter AF, Cook IA, Gilmer WS, Marangell LB, Burgoyne KS, Howland RH, Trivedi MH, Zisook S, Jain R, Fava M, Iosifescu D, Greenwald S. Effectiveness of a quantitative electroencephalographic biomarker for predicting differential response or remission with escitalopram and bupropion in major depressive disorder. Psychiatry Res. 2009 Sep 30;169(2):132-8. doi: 10.1016/j.psychres.2009.04.004. Epub 2009 Aug 26. PMID 19709754
- [Derived] Cook IA, Hunter AM, Gilmer WS, Iosifescu DV, Zisook S, Burgoyne KS, Howland RH, Trivedi MH, Jain R, Greenwald S, Leuchter AF. Quantitative electroencephalogram biomarkers for predicting likelihood and speed of achieving sustained remission in major depression: a report from the biomarkers for rapid identification of treatment effectiveness in major depression (BRITE-MD) trial. J Clin Psychiatry. 2013 Jan;74(1):51-6. doi: 10.4088/JCP.10m06813. PMID 23419226